CLINICAL TRIAL: NCT06725797
Title: Pilot Study on the Effectiveness of Sulphurous Thermal Water in Wound Hygiene: Spa Wound Care
Brief Title: Study on the Effectiveness of Hypothermal Sulphurous Water in Wound Hygiene
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Università degli studi di Roma Foro Italico (Other)
Responsible Party: Principal Investigator, Mario Fontana, MD, PhD, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VULNOLOGIATERMALE1; AR12419075FF92A2 (Other Grant/Funding Number: La Sapienza University of Rome)
Record Dates: First submitted 2024-11-11; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Ulcers; Wound - in Medical Care; Wounds and Injuries; Wound Healing; Wound Care; Venous Ulcers; Wound Cleansing
Keywords: wound hygiene; chronic wound; sulfurous water; spa thermal water; wound care
MeSH Terms: conditions — Ulcer; Wounds and Injuries; Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: The study is an interventional pilot trial assessing the efficacy of hypothermal sulphurous thermal water (STW) in the wound hygiene of patients affected by hard to heal, chronic, infected wounds. The eligible subjects will be 1:1 randomized in two arms and treated with pure sulfurous spa water, already authorized for medical drinking therapy, on soaked gauzes (GROUP A) or for full limb immersion (GROUP B) for 20 minutes. Ph, Trans epidermal water loss (TEWL), healing rate (Bates-Jensen Wound Assessment Tool) wound fluorescence imaging for bacterial colonization and wound microbiome will be tested at 3 timepoints: T0 (prior treatment), T1 (just after treatment) , Tf (complete wound re-epithelization).
Who Masked: Outcomes Assessor
Masking Description: Microbiological and microbiome assessors are blinded to subjects' treatment or arm randomization list.
  Epidemiological and statistic assessors are blinded to arm randomization list as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A:wound hygiene with spa thermal sulphurous water delivered with pack on soaked gauzes (Active Comparator): non woven gauzes will be soaked with sulphurous thermal water and positioned on the wound as packs for 20 minutes, at spring temperature (23°C).
  Interventions: Procedure: wound hygiene with hypothermal sulfurous water by packs
- GROUP B: limb full immersion in spa thermal sulphurous water (Active Comparator): full wound immersion: the limb hosting the wound is located in a limb-sized tube filled with sulphurous water for 20 minutes at spring temperature (23°C).
  Interventions: Procedure: wound hygiene with hypothermal sulfurous water by limb full immersion

INTERVENTIONS:
Procedure: wound hygiene with hypothermal sulfurous water by packs — GROUP A: After dressing removal, the wound is exposed. Sulphur thermal water at spring temperature (23°C) is applied for 20 minutes on the untreated wound by packs on non woven gauzes entirely covering the area. Eventually, if dried, gauzes are externally watered with additional sulphurous thermal water during the 20 minutes. After water application the wound follows the other 3 steps of the wound hygiene protocol: non viable tissue removal, edges reactivation and dressing. Non interactive dressings, just for wound moisture management, are used on cleaned wound/s. Dressing fixation, elastic bandages or off-load will be provided when required. the intervention will be repeated every 48 hours for both arms.
  Other Names: wound hygiene by packs
  Arms: GROUP A:wound hygiene with spa thermal sulphurous water delivered with pack on soaked gauzes
Procedure: wound hygiene with hypothermal sulfurous water by limb full immersion — GROUP B: After dressing removal, the wound is exposed. Sulphur thermal water at spring temperature (23°C) is applied for 20 minutes on the untreated wound by limb full immersion in a limb tub. After the immersion, the wound follows the other 3 steps of the wound hygiene protocol: non viable tissue removal, edges reactivation and dressing. Non interactive dressings, just for wound moisture management, are used on cleaned wound/s. Dressing fixation, elastic bandages or off-load will be provided when required. the intervention will be repeated every 48 hours for both arms.
  Other Names: wound hygiene by limb full immersion
  Arms: GROUP B: limb full immersion in spa thermal sulphurous water

SUMMARY:
This is an interventional double arms pilot study on the effectiveness of hydrogen sulfide (H2S) rich and microbiologically pure spa sulphurous water, in the wound hygiene of hard-to heal wounds, set in an italian spa facility. At least 24 subjects enrolled according to selection criteria will be 1:1 randomized in two intervention groups: the former (A) undergoing pack of sulphurous water on soaked gauzes for 20 minutes, the latter (B) undergoing full limb immersion for 20 minutes. Differences among the two arms will be assessed as changes in wound microbiome, wound pH, Trans epidermal water loss (TEWL), 1000x ex-vivo microscope imaging, wound fluorescence imaging for bacterial colonization and longitudinal shifts in wound sizing and peculiar features according to the Bates-Jensen Wound Assessment Tool (BWAT). Time required for re-epithelization will be recorded together with any adverse reactions or events for both arms and compared. The study aims at assessing the effectiveness of hydrogen sulfide exogenous supply on infected or colonized hard to heal wounds and which way of administration (pack Vs immersion) could have prevailing effects.

DETAILED DESCRIPTION:
The effectiveness of sulphurous thermal waters in the treatment of complex or difficult wounds has been known since ancient times.

In recent years, the increase in life expectancy, the aging of the population and survival of chronically ill subjects lead to the outbreak of "hard to heal" wounds presenting multi drug resistant germs (MDR). Recent studies have shown that the effectiveness of thermal waters is not only related to the presence of dissolved ions but, as in the case of sulphurous ones, to the presence of hydrogen sulfide, a gas transmitter that diffuses freely through the skin, eliciting local and systemic effects. This molecule, present in sulphurous waters within specific pH and temperature ranges, is able to promote the healing of acute, chronic and infected wounds. H2S also exerts a powerful antibacterial and antifungal effect by transforming into pentationic acid (H2S5O6). In addition, the specific microbiome of each thermal source has the ability to interact with the skin microbiome and prevails over wound biofilm stimulating skin eubiosis. By virtue of these considerations, investigators perform an interventional pilot trial conducted to evaluate the effects of raw sulphurous thermal water, microbiologically pure, in the wound hygiene of acute and chronic wounds, regardless of their aetiology and bacterial colonization.

Outpatients >18 years, presenting at spa facility with wound respecting selection criteria, will undergo to a wound hygiene protocol based on the use of raw sulphurous thermal water of Acque Albule, tested negative to microbiological analysis for the presence of pathogens. Subjects will be 1:1 randomized in 2 treatment arms: group A receiving sulphurous thermal water pack on soaked gauzes for 20 minutes and group B having their wound/s fully immersed in sulphurous thermal water for 20 minutes. Both arms will be treated every 48 hours up to complete wound re-epithelization. Participants will be submitted just at enrollment to wound microbiological sampling (swab). All parameters worth investigating will be assessed at each session prior to intervention (T0,2,4..) and after (T1,3,5…). Specifically wound microbiome sampling, together with pH, trans epidermal water loss (TEWL) measurements, wound fluorescence bacterial imaging, and ex-vivo microscope imaging will be recorded at each time point. Any adverse events, superinfections will be monitored and properly managed. A three months post-healing follow-up (Tf) will be performed to determine scar quality and possible wound relapse. Results will be expressed in term of intra-session (short term effects) and inter sessions(longitudinal effects) changes (delta) in order to assess the singular and the whole effects of each arm intervention. Finally differences in term of effectiveness among the two interventions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Any comorbidities (except very severe I, II immune deficiencies)
* Any systemic drug therapy
* Any associated dressing (except peroxides)
* Acute or chronic wounds requiring wound care treatment
* Genital/oral wounds
* Infected wounds, including MDR pathogens
* Biofilmed wounds

Exclusion Criteria:

* Unexplored fistula
* Enteric fistula
* Exposure of fascia, vessels, bones, organs
* Pyoderma Gangrenosum (monotherapy)
* Implanted or penetrating devices (CVC , Port-a-cath, drainages, peritoneal dialysis, external fixators....etc.)
* Exposed implants(nails, plates, internal defibrillator, Pace maker)
* Local antibiotic therapy (not supported by antibiogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
wound healing rate | within 10 minutes after wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  Longitudinal Wound healing rate will be assessed at each dressing change by applying Bates Jansen Wound Tool Score (BWAT)., max score 65, min 13, The HIGHER the total score, the more severe the wound status.
Short term Wound bacteria critical colonization | within 10 minutes before wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  The fluorescence wound imaging using Moleculight device, assessing critical bacterial colonization (>104UFC) of the wound before intervention will be compared to that obtained after intervention to determine whether 20 minutes exposure to sulphurous water could have exerted an antibacterial activity. The HIGHER the luminescence, the more severe the wound critical colonization
Short term Wound microbiome changes | within 10 minutes before and within 10 minutes after wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  Wound microbiome changes will be determined before treatment, immediately after the wound hygiene in order to assess its variation related to sulfurous hypothermal water exposure .(analysis of 16S ribosomial rNa sub-unit)
Short Term Wound bed pH changes | within 10 minutes before and within 10 minutes after wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  Ph of the wound bed will be measured using a flat glass cleavable probe, before and after intervention in order to detect if 20 minutes exposure to soaked gauzes in H2S rich water are enough to determine a lowering in wound pH values.(according to pH scale 0 to 10)

SECONDARY OUTCOMES:
Longitudinal Wound microbiome changes during treatment up to re-epithelization | within 10 minutes before wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  Wound microbiome changes will be determined comparing samples collected before intervention every 48 hours in order to assess inter sessions quantitative and qualitative changes related to sulfurous hypothermal water exposure (analysis of 16S risosomial rNA sub-units).
Longitudinal Wound bacterial critical colonization control | within 10 minutes before wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  Referring to the microbiological swab performed at enrollment on day 0, The fluorescence wound imaging using Moleculight device,will monitor any eventual inter session changes in critical bacterial colonization of the wound up to re-epithelization.The HIGHER the total wound luminescence, the more severe the wound bacterial colonization.
Longitudinal Wound bed pH changes | within 10 minutes before wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  Ph of the wound bed, measured using a flat glass cleavable probe, at each session , before the exposure to H2S rich water are compared in order to assess an inter session lowering trend of wound pH (pH scale from 0 to 10).
Longitudinal Wound TEWL changes | within 10 minutes before wound hygiene, each session, every 48 hours, from day 0 up to wound re-epithelialization (up to 1 year)
  TEWL (TRANS EPIDERMAL WATER LOSS) of the wounded skin will be measured in g hm -2 ,using a closed chamber device, at each session, before the intervention. The inter session values obtained will be compared to assess an eventual lowering trend of TEWL values, a sign of recovery of skin integrity typically associated to wound re-epithelization . Normal values are considered ranging from 0 to 15 g hm -2 ). The HIGHER the TEWL score, the more severe the skin breakdown
Long term re-epithelization stability | 90 days after wound healing (Tf)
  Wound area integrity and neo-epithelium stability (by skin plication manoeuvre) are evaluated 90 days after complete wound healing together with any wound relapse (physical examination: presence Vs absence).

OTHER OUTCOMES:
Microbiological wound sampling | at enrollment, day 0
  A swab for microbiological identification of wound colonizing pathogens will be collected at enrollment. The swab will likely identify bacteria species, + CFU (colony forming Units) or the strength of bacterial colonization.
Effects of H2S rich water on wound biofilm integrity | within 10 minutes before and within 10 minutes after wound hygiene, each session, every 48 hours from day 0 up to wound re-epithelialization (up to 1 year)
  Using an in vivo 1000x bluetooth microscope, the details of biofilm appearance/integrity will be compared both in short term and longitudinally. The HIGHER the biofilm appearance, the more severe the wound chronicity.
Short term differences among the two arms: administration of H2S could impact on the effectiveness of re-epithelization | within 10 minutes before and within 10 minutes after wound hygiene, each session, every 48 hours from day 0 up to wound re-epithelialization (up to 1 year)
  The whole Intra sessions parameters (BWAT score, pH, TEWL, fluorescence bacterial load), results obtained in both arms will be compared in order to assess any differences among the two way of administrations and which one might have prevailing effects.(p value)
Longitudinal differences among the two arms | within 10 minutes before wound hygiene, each session, every 48 hours from day 0 up to wound re-epithelialization (up to 1 year)
  The whole Inter sessions parameters results (BWAT score, pH, TEWL, days for negativization of bacterial colonization, days to complete reepithelization), obtained in both arms will be compared in order to assess any differences among the two way of administrations and which one might have prevailing effects.(p value)

CONTACTS AND LOCATIONS:
Overall Officials: Serena Crucianelli, MD, Principal Investigator — La Sapienza University of Rome; Mario Fontana, MD, PhD, Study Director — La Sapienza University of Rome; Vincenzo Romano Spica, MD, PhD, Study Chair — Foro Italico University of Rome
Locations (1):
- Terme di Roma Acque Albiule, Bagni di Tivoli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
raw data not containing any tracking sensible data (whole data) will be shared for publishing and at authorized medical conferences

REFERENCES:
- [Background] Tsuji, Hideo.
- [Background] Faga A, Nicoletti G, Gregotti C, Finotti V, Nitto A, Gioglio L. Effects of thermal water on skin regeneration. Int J Mol Med. 2012 May;29(5):732-40. doi: 10.3892/ijmm.2012.917. Epub 2012 Feb 15. PMID 22344563
- [Background] Davidelli S, Bassetto F, Vitale M, Scapagnini G. Thermal Waters and the hormetic effects of hydrogen Sulfide on inflammatory arthritis and wound healing. Chapter 10 elsevier https://www.sciencedirect.com/science/article/pii/B9780128142530000103
- [Background] Wallace JL, Dicay M, McKnight W, Martin GR. Hydrogen sulfide enhances ulcer healing in rats. FASEB J. 2007 Dec;21(14):4070-6. doi: 10.1096/fj.07-8669com. Epub 2007 Jul 18. PMID 17634391
- [Background] Mormile I, Tuccillo F, Della Casa F, D'Aiuto V, Montuori N, De Rosa M, Napolitano F, de Paulis A, Rossi FW. The Benefits of Water from Nitrodi's Spring: The In Vitro Studies Leading the Potential Clinical Applications. Int J Mol Sci. 2023 Sep 5;24(18):13685. doi: 10.3390/ijms241813685. PMID 37761993
- [Background] Napolitano F, Postiglione L, Mormile I, Barrella V, de Paulis A, Montuori N, Rossi FW. Water from Nitrodi's Spring Induces Dermal Fibroblast and Keratinocyte Activation, Thus Promoting Wound Repair in the Skin: An In Vitro Study. Int J Mol Sci. 2023 Mar 10;24(6):5357. doi: 10.3390/ijms24065357. PMID 36982430
- [Background] Ahmad A, Druzhyna N, Szabo C. Effect of 3-mercaptopyruvate Sulfurtransferase Deficiency on the Development of Multiorgan Failure, Inflammation, and Wound Healing in Mice Subjected to Burn Injury. J Burn Care Res. 2019 Feb 20;40(2):148-156. doi: 10.1093/jbcr/irz007. PMID 30649358
- [Background] Benedetti F, Curreli S, Krishnan S, Davinelli S, Cocchi F, Scapagnini G, Gallo RC, Zella D. Anti-inflammatory effects of H2S during acute bacterial infection: a review. J Transl Med. 2017 May 10;15(1):100. doi: 10.1186/s12967-017-1206-8. PMID 28490346
- [Background] Sheng L, Zhang Z, Zhang Y, Wang E, Ma B, Xu Q, Ma L, Zhang M, Pei G, Chang J. A novel "hot spring"-mimetic hydrogel with excellent angiogenic properties for chronic wound healing. Biomaterials. 2021 Jan;264:120414. doi: 10.1016/j.biomaterials.2020.120414. Epub 2020 Sep 19. PMID 32980635
- [Background] Han X, Wang L, Shang Y, Liu X, Yuan J, Shen J. Hydrogen sulfide-releasing polyurethane/gelatin/keratin-TA conjugate mats for wound healing. J Mater Chem B. 2022 Nov 3;10(42):8672-8683. doi: 10.1039/d2tb01700h. PMID 36250498
- [Background] Wu J, Chen A, Zhou Y, Zheng S, Yang Y, An Y, Xu K, He H, Kang J, Luckanagul JA, Xian M, Xiao J, Wang Q. Novel H2S-Releasing hydrogel for wound repair via in situ polarization of M2 macrophages. Biomaterials. 2019 Nov;222:119398. doi: 10.1016/j.biomaterials.2019.119398. Epub 2019 Aug 16. PMID 31487582
- [Background] Wu J, Li Y, He C, Kang J, Ye J, Xiao Z, Zhu J, Chen A, Feng S, Li X, Xiao J, Xian M, Wang Q. Novel H2S Releasing Nanofibrous Coating for In Vivo Dermal Wound Regeneration. ACS Appl Mater Interfaces. 2016 Oct 19;8(41):27474-27481. doi: 10.1021/acsami.6b06466. Epub 2016 Oct 7. PMID 27504858
- [Background] Zhang Y, Yue T, Gu W, Liu A, Cheng M, Zheng H, Bao D, Li F, Piao JG. pH-responsive hierarchical H2S-releasing nano-disinfectant with deep-penetrating and anti-inflammatory properties for synergistically enhanced eradication of bacterial biofilms and wound infection. J Nanobiotechnology. 2022 Jan 29;20(1):55. doi: 10.1186/s12951-022-01262-7. PMID 35093073
- [Background] Cremonini, V., Giuliani, R., Fusaroli, P., & Rubbi, I. Valutazione e monitoraggio delle ferite difficili con l'utilizzo della scala Bates-Jensen Assessment Tool: studio osservazionale. - DERMATOLOGICAL EXPERIENCES 2017;19:1-2. DOI: 10.23736/S1128-9155.17.00446-0
- [Background] Pinnagoda J, Tupker RA, Agner T, Serup J. Guidelines for transepidermal water loss (TEWL) measurement. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1990 Mar;22(3):164-78. doi: 10.1111/j.1600-0536.1990.tb01553.x. PMID 2335090
- [Background] Schneider LA, Korber A, Grabbe S, Dissemond J. Influence of pH on wound-healing: a new perspective for wound-therapy? Arch Dermatol Res. 2007 Feb;298(9):413-20. doi: 10.1007/s00403-006-0713-x. Epub 2006 Nov 8. PMID 17091276
- [Background] Wilson IA, Henry M, Quill RD, Byrne PJ. The pH of varicose ulcer surfaces and its relationship to healing. Vasa. 1979;8(4):339-42. No abstract available. PMID 44410
- [Background] Toriyama T, Kumada Y, Matsubara T, Murata A, Ogino A, Hayashi H, Nakashima H, Takahashi H, Matsuo H, Kawahara H. Effect of artificial carbon dioxide foot bathing on critical limb ischemia (Fontaine IV) in peripheral arterial disease patients. Int Angiol. 2002 Dec;21(4):367-73. PMID 12518118
- [Background] Zhao H, Lu S, Chai J, Zhang Y, Ma X, Chen J, Guan Q, Wan M, Liu Y. Hydrogen sulfide improves diabetic wound healing in ob/ob mice via attenuating inflammation. J Diabetes Complications. 2017 Sep;31(9):1363-1369. doi: 10.1016/j.jdiacomp.2017.06.011. Epub 2017 Jun 30. PMID 28720320
- [Result] Crucianelli, S., Fontana, M., Moretti, F., Cocomello, N., Mariano, A., & DEL BEN, M. (2024). PILOT STUDY ON THE EFFECTIVENESS OF SULFUROUS THERMAL WATER IN WOUND HYGIENE: SPA WOUND CARE. In The 24th Annual Meeting of the European Pressure Ulcer Advisory Panel Abstract book (pp. 81-81).

DOCUMENTS (1):
  • Informed Consent Form (2024-10-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT06725797/ICF_000.pdf